CLINICAL TRIAL: NCT02002182
Title: Window of Opportunity Trial of Neoadjuvant ADXS 11-001 Vaccination Prior to Robot -Assisted Resection of HPV-Positive Oropharyngeal Squamous Cell Carcinoma
Brief Title: ADXS 11-001 Vaccination Prior to Robotic Surgery, HPV-Positive Oropharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Sikora (Other)
Collaborators: Advaxis, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Andrew Sikora, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-36001 GCO 13-1411
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of the Head and Neck; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: HPV; oropharynx; squamous cell carcinoma; head and neck cancer; transoral robotic surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment-Vaccine Group (Experimental): Two vaccinations with ADXS11-001 (ADXS-HPV) will be given at a dose of 1x10^9 cfu intravenously. The drug will be given as a 500ml infusion over 60 minutes.
  Interventions: Biological: ADXS11-001 (ADXS-HPV)
- Control Group (No Intervention): Observational control group treated with standard of care therapy only

INTERVENTIONS:
Biological: ADXS11-001 (ADXS-HPV) — ADXS11-001 (ADXS-HPV) is a live attenuated Listeria monocytogenes (Lm)-LLO immunotherapy developed for the treatment of HPV-associated dysplasia and malignancy.
  Other Names: ADXS11-001; ADXS-HPV
  Arms: Treatment-Vaccine Group

SUMMARY:
Some cancers may be related to an infection with a virus, such as the Human Papilloma Virus (HPV). HPV related Oropharyngeal cancer (HPVOPC) accounts for 80% of oropharynx cancer cases in the United States. HPVOPC has better prognosis than patients with HPV negative oropharynx cancer. In many hospitals, the standard of care treatment for oropharyngeal cancer is surgery and/or radiotherapy with or without chemotherapy. While chances of survival for most patients with HPVOPC is very good, current treatments are associated with short- and long-term side effects which can be severe. In pre-clinical research using animal models of cancer, vaccination targeting the HPV virus has been found to cause tumor regression. Thus, approaches which target the unique characteristics of HPV-infected cancer cells, such as therapeutic vaccination, are attractive strategies for potentially reducing radiotherapy and chemo radiotherapy regimens (and thus decreasing toxicity) and enhancing long-term disease control.

The purpose of this study is to see if an experimental vaccine, ADXS11-001, is effective in stimulating the body's defense system against HPV-positive oropharyngeal squamous cell carcinoma before transoral (through the mouth) surgery. The experimental product ADXS11-001 uses a live strain of the Listeria monocytogenes (Lm) bacteria that has been genetically modified such that the risk of getting an infection is significantly reduced. Several research studies have already been conducted with ADXS11-001 in men and women with cancer. So far, approximately 722 doses of ADXS11-001 have been given to 290 patients with HPV associated cancers.

DETAILED DESCRIPTION:
This is an investigator-initiated prospective clinical study of patients with stage I-IV squamous cell carcinoma of the oropharynx (OPSCC) who are to undergo ablative transoral robotic surgery (TORS).

There is a vaccination group and a control group in this study.

Subjects in the control group will not receive the vaccination and will only be followed after TORS surgery for additional research blood tests to measure how their immune system is working.

Subjects in the vaccination group will receive two vaccinations prior to surgery. The first dose will be about 33 days before surgery, and the second will be about 14 days before surgery.

Participation in this study will also include allowing the research team to take several blood samples from the subject at various times before, during, and after treatment for his/her cancer.

Vaccination subjects will be monitored closely after treatment and includes 6 months of oral antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* The patient has newly-diagnosed, biopsy proven squamous cell carcinoma of Stage I-IV (T1-3, N0-2b) of the oropharynx.
* The patient's tumor is HPV positive by PCR or ISH assay of tumor biopsy.
* The patient is able/eligible to undergo treatment with transoral robotic surgery (TORS) with or without neck dissection and with or without adjuvant radiation therapy or chemoradiation.
* The patient is able to understand and give informed consent.
* The patient is at least 18 years old.
* The patient's ECOG performance status is </= 2.

Exclusion Criteria:

* The patient has had prior head and neck squamous cell carcinoma (HNSCC), with the exception of superficial cutaneous basal cell or squamous cell carcinomas.
* The patient has active cancer in another part of the body, with the exception of superficial cutaneous basal cell or squamous cell carcinomas
* If a cancer survivor, the disease free interval is less than 3 years, with the exception of superficial cutaneous basal cell or squamous cell carcinomas.
* If a cancer survivor the patient received prior systemic chemotherapy or radiotherapy
* If prior standard-of-care pre-treatment biopsy is inadequate for analysis by immunohistochemistry, and the patient is unwilling to undergo an additional biopsy procedure.
* The patient is a prisoner.
* The patient has a psychiatric illness or developmental delay which would interfere with understanding of the study and provision of informed consent.
* The patient has previously received definitive surgical, radiation, or chemoradiation treatment for HNSCC.
* The patient has a history of HIV or other known cause of immunosuppression, or is actively taking immunosuppressive medications due to organ transplantation, rheumatoid disease, or other medical conditions.
* Patient is allergic to naproxen or Ibuprofen.
* The patient has a history of liver disease.
* The patient has a contraindication (e.g. sensitivity/allergy) to both trimethoprim/sulfamethoxazole and ampicillin.
* The patient has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)). NOTE: More common devices and prosthetics which include arterial and venous stents, dental and breast implants and venous access devices (e.g. Port-a-Cath or Mediport) are permitted.
* Patients who are receiving or may receive future treatment with PI3K or TNFα inhibitors.
* Patients who have undergone a major surgery, including surgery for a new artificial implant and/or device, within 6 weeks prior to the initiation of ADXS11-001 treatment. Sponsor must be consulted prior to enrolling subjects on the study who recently had a major surgery or have new artificial implant, and/or devices.
* Patients who have a history of listeriosis or prior ADXS11-001 therapy.
* Patients with a known allergy to any component of the study treatment formulations.
* Pregnancy. The effects of this vaccine on the developing human fetus are unknown. For this reason women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2018-07-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Sikora, MD PhD, Study Chair — Baylor College of Medicine; Brett Miles, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment-Vaccine Group | Control Group
Started | 9 | 6
Completed | 4 | 5
Not Completed | 5 | 1
Not completed — Withdraw from study | 3 | 1
Not completed — Health Reasons | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Vaccine Group | Control Group | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Median (Full Range); unit: years] | 72 [51 to 91] | 53 [49 to 62] | 62 [49 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: HPV-Specific T Cell Response Rate
Description: Response rate defined as proportion of participants with a >2-fold increase in HPV-specific T cell response from baseline to time of surgery.
Time Frame: At time of surgery
Population: The analysis included participants who had HPV-specific T cell response measurement at time of surgery. T cell response data were not collected at time of surgery for the control group, which was an optional observational group.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment-Vaccine Group | Control Group
Number analyzed (Participants) | 9 | 0
proportion of participants | 0.333 [0.075 to 0.701] |

2. Primary Outcome: Number of Participants With Any Grade 3 or 4 Toxicity
Description: Degree of toxicity assessed according to NCI Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria.
Time Frame: Assessed up to 30 Days after surgery
Population: All participants were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Vaccine Group | Control Group
Number analyzed (Participants) | 9 | 6
Participants | 5 | 1

3. Secondary Outcome: HPV-Specific T Cell Response Rate
Description: Response rate defined as proportion of participants with a >2-fold increase in HPV-specific T cell response from baseline to 3 months after surgery.
Time Frame: Assessed up to 3 months after surgery
Population: The analysis included participants who had at least one HPV-specific T cell response measurement post surgery.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment-Vaccine Group | Control Group
Number analyzed (Participants) | 8 | 4
proportion of participants | 0.625 [0.245 to 0.915] | 0.75 [0.194 to 0.994]

ADVERSE EVENTS:
Time Frame: Up to 3 year post treatment for the vaccinated group or post surgery for the control group.
Description: Adverse events (AE) were collected starting on the first day of vaccine administration and evaluated for severity and relationship to treatment for 30 days post treatment and for 3 year safety observation period. AE of grade 3 or higher were designated severe adverse events (SAE).
Arm/Group | Treatment-Vaccine Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/9 | 1/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-Vaccine Group (N=9) | Control Group (N=6)
Hypertension (Cardiac disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Failure to thrive (General disorders) | 1 (1) | 0 (0)
Mouth pain (General disorders) | 0 (0) | 1 (1)
Pain in throat and left ear when swollowing (General disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
mucositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-Vaccine Group (N=9) | Control Group (N=6)
Decreased WBCs (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Localized edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
lymphedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (HR112) (Cardiac disorders) | 1 (1) | 0 (0)
Tachychardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Face Flushing (Endocrine disorders) | 1 (1) | 0 (0)
Flushed Face (Endocrine disorders) | 1 (1) | 0 (0)
Flushing (Endocrine disorders) | 2 (2) | 0 (0)
Flushing (face+neck) (Endocrine disorders) | 1 (1) | 0 (0)
Sweating (Endocrine disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Difficulty with swallowing solid food (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 7 (12) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intermittent diarrhea after taking Bactrim (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (7) | 2 (2)
Upset Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
tongue ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia (General disorders) | 3 (3) | 0 (0)
Body ache (General disorders) | 3 (3) | 0 (0)
Chill (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 7 (10) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 2 (2)
Ear pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (8) | 1 (1)
Fever (General disorders) | 5 (7) | 0 (0)
Intermittent throat pain when swallowing (General disorders) | 1 (2) | 0 (0)
Jaw pain (General disorders) | 0 (0) | 1 (1)
Left Ear Pain (General disorders) | 0 (0) | 1 (1)
Mild discomfort in the throat on the left side (General disorders) | 1 (1) | 0 (0)
Mild odynophagia (General disorders) | 0 (0) | 1 (1)
Mild throat pain (General disorders) | 0 (0) | 1 (1)
Neck Mass (General disorders) | 0 (0) | 1 (1)
Occasional fatigue (General disorders) | 1 (1) | 0 (0)
Occasional pain in throat (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (3)
Pain (in neck) (General disorders) | 0 (0) | 1 (1)
Pain (in throat) (General disorders) | 0 (0) | 1 (1)
Pain in left jaw (General disorders) | 1 (1) | 0 (0)
Pain in legs (General disorders) | 1 (1) | 0 (0)
Pain in neck (General disorders) | 0 (0) | 1 (1)
Pain in right ear (General disorders) | 1 (1) | 0 (0)
Pain in right ear,nec (General disorders) | 1 (1) | 0 (0)
Pain in right shoulder (General disorders) | 1 (1) | 1 (2)
Pain in right side of neck (General disorders) | 0 (0) | 1 (1)
Right Neck Pain (General disorders) | 0 (0) | 1 (1)
Right Shoulder Pain (General disorders) | 1 (1) | 0 (0)
Shivering (General disorders) | 1 (2) | 0 (0)
Slight sore throat (General disorders) | 1 (1) | 0 (0)
Throat pain (General disorders) | 2 (2) | 0 (0)
Tonsillar Pain (General disorders) | 0 (0) | 1 (1)
Weakening (General disorders) | 1 (1) | 0 (0)
Xerostomia (General disorders) | 1 (1) | 1 (1)
dry saliva (General disorders) | 0 (0) | 1 (1)
left buccal mucosa lump (General disorders) | 0 (0) | 1 (1)
minor discomfort when swallowing (General disorders) | 1 (1) | 0 (0)
pain in right neck (General disorders) | 1 (1) | 0 (0)
pain in right neck, shoulder (General disorders) | 1 (1) | 0 (0)
pain in shoulder (General disorders) | 0 (0) | 1 (1)
pain in throat (General disorders) | 3 (5) | 0 (0)
pressure in the right neck (General disorders) | 0 (0) | 1 (1)
slight tightness on outside of left neck at surgical site when out in the cold only (General disorders) | 1 (1) | 0 (0)
tooth decay (General disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intermittent neck stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cramping in feet (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Decreased taste (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 0 (0)
Headache Intermittent (Nervous system disorders) | 1 (1) | 0 (0)
Loss of taste (Nervous system disorders) | 0 (0) | 1 (2)
Memory loss and cognitive decline (Nervous system disorders) | 1 (1) | 0 (0)
Numbness right Ear,Neck and back of head (Nervous system disorders) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Blood tinged sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Voice Change (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
voice changes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mucositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (chest, back of neck) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
left lump posterior pharyngeal region (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
radiation associated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
tender left arm lump (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02002182/Prot_SAP_000.pdf